CLINICAL TRIAL: NCT00711672
Title: Critical Negotiations: Narrative Agreement, Negotiation, and Register Use in Encounters Between Patients With Metastatic Colorectal Carcinoma and Their Oncologists
Brief Title: Study of the Therapeutic Use of Language in Patients With Metastatic Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Hematology and Oncology Associates of NE Pennsylvania (Other)
Responsible Party: Christian S Adonizio MD, Hematology and Oncology Associates of Northeastern Pennsylvania, PC
Other Study IDs: 808231
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2011-06

CONDITIONS: Colorectal Cancer
Keywords: Personal Communication; Doctor Patient Relations; Narrative Medicine
MeSH Terms: conditions — Colorectal Neoplasms; Communication; Narrative Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Medical Oncologists treating patients with metastatic colorectal cancer
- 2: Patients with metastatic colorectal cancer receiving re-staging CT scans

SUMMARY:
The purpose of this study is to determine if the degree of agreement between patients and their physicians regarding the "story" of the illness correlates with improved patient symptom control and quality of life. Another goal of the study is to examine the actual language used by patients and physicians in a specific clinical situation.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the co-created therapeutic narrative in scheduled office visits between adult patients with metastatic colorectal carcinoma and their medical oncologists in a community practice setting. The study will focus on the negotiation of the illness narrative and the semiotic (primarily linguistic) tools employed. The study will involve patients from a large community cancer center from Northeastern Pennsylvania (this center sees about 3,000 new patients each year). About 85% of patients with cancer in the United States are treated in this type of setting (National Cancer Institute, 2007), and so many results from this population are applicable to most cancer patients in the United States. The location of this study makes it very different from the majority of medical anthropological studies that are usually performed in urban academic medical centers or in sites outside of the United States or Western Europe. Although community cancer centers are the location of most of the treatment of patients with cancer in the United States, there are few to no studies published studying this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients and Physicians at Hematology and Oncology Associates of NE Pennsylvania
* Patients must have metastatic (stage IV) colorectal carcinoma
* Patients must be on treatment for their disease
* Patients must be scheduled for re-staging CT scans
* Patients must be older than 18 years old

Exclusion Criteria:

* Patients with a diagnosis other than metastatic colorectal carcinoma
* Patients not receiving active treatment or not having re-staging CT scans
* Patients younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal carcinoma and their physicians at a large community cancer center in Northeastern Pennsylvania.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Correlation of degree of "narrative agreement" with validated quality of life measures | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Adonizio, MD, Principal Investigator — Hematology and Oncology Associates of NE Pennsylvania
Locations (1):
- Hematology and Oncology Associates of Northeastern Pennsylvania, PC, Dunmore, Pennsylvania, United States

REFERENCES:
- [Background] Agha, A. (2007). Language and Social Relations. Studies in the Social and Cultural Foundations of Language. Cambridge, Cambridge University Press. 24: 242-244.
- [Background] Ainsworth-Vaughn, N. (1998). Claiming Power in Doctor-Patient Talk. New York, Oxford University Press.
- [Background] Austin, J.L. (1975) How to do things with Words. Ed. J.O. Urmson and Marina Sbisa. Cambridge, MA, Harvard University Press.
- [Background] Briggs, C. (1986) Learning How to Ask:A sociolinguistic appraisal of the role of the interview in social science research. Cambridge, Cambridge University Press.
- [Background] Cassel EJ. The nature of suffering and the goals of medicine. N Engl J Med. 1982 Mar 18;306(11):639-45. doi: 10.1056/NEJM198203183061104. PMID 7057823
- [Background] Cassell, E. J. (1991). The Nature of Suffering and the Goals of Medicine. New York, Oxford University Press: 37-43.
- [Background] Charon, R. (2006). Narrative Medicine: Honoring the Stories of Illness. New York, Oxford.
- [Background] Csordas, T. J. ed. (1994). Embodiment and experience: The existential ground of culture and self. Cambridge Studies in Medical Anthropology. Cambridge: Cambridge University Press.
- [Background] Gee, J.P. (2005) An Introduction to Discourse Analysis: Theory and Method, 2nd ed. New York, Routledge.
- [Background] Eggly S. Physician-patient co-construction of illness narratives in the medical interview. Health Commun. 2002;14(3):339-60. doi: 10.1207/S15327027HC1403_3. PMID 12186492
- [Background] Ferrell BR, Dow KH, Grant M. Measurement of the quality of life in cancer survivors. Qual Life Res. 1995 Dec;4(6):523-31. doi: 10.1007/BF00634747. PMID 8556012
- [Background] Foucault, M. (1994). The Birth of the Clinic: An Archaeology of Medical Perception. New York, NY, Vintage Books.
- [Background] Frank, A. W. (1995). The Wounded Storyteller: Body, Illness, and Ethics. Chicago, Chicago University Press.
- [Background] Goffman, E. (1963) Stigma: Notes on the Management of Spoiled Identity. Englewood Cliffs, Prentice Hall.
- [Background] Good, B. J. (1994). Medicine, Rationality, and Experience: an anthropological perspective. Cambridge, Cambridge University Press.
- [Background] Laderman, C. and M, Roseman eds (1996) The Performance of Healing. London, Routledge.
- [Background] Linde, C. (1993) Life Stories: The Creation of Coherence. New York, Oxford University Press.
- [Background] Lock, M. and N. Scheper-Hughes (1996). A Critical-Interpretive Approach in Medical Anthropology: Rituals and Routines of Discipline and Dissent. Medical Anthropology: Contemporary Theory and Method. C. F. Sargent and T. M. Johnson. Westport, CT, Praeger Publishers: 47.
- [Background] Lyotard, J.-F. (1984). The Postmodern Condition: A Report on Knowledge. Minneapolis, University of Minnesota Press.
- [Background] Lortie F. Healing dramas and clinical plots: the narrative structure of experience. BMJ. 1999 May 1;318(7192):1219. doi: 10.1136/bmj.318.7192.1219. No abstract available. PMID 10221969
- [Background] Mehan, H. (1996). The Construction of an LD student: A case study in the politics of Representation. Natural Histories of Discourse. M. Silverstein and G. Urban. Chicago, The University of Chicago Press: 253-276.
- [Background] Mishler, E. G. (1984). The Discourse of Medicine: Dialectics of Medical Interviews. Norwood, NJ, Ablex Publishing Corporation.
- [Background] National Cancer Institute (2007). "NCI Community Cancer Centers Program Pilot 2007-2010." from http://ncccp.cancer.gov/Media/FactSheet.htm.
- [Background] Riessman, Catherine Kohler. (1993) Narrative Analysis. Newbury Park, Sage University Paperback
- [Background] Ross, N. (2004). Culture and Cognition: Implications for Theory and Method. Thousand Oaks, CA, Sage
- [Background] Sontag, S. (2002). Illness as Metaphor and AIDS and Its Metaphors. New York, Penguin Books.
- [Background] The University of Texas--M.D.Anderson Cancer Center. (1999) "MDASI, M.D. Anderson Symptom Inventory Core Items", University of Texas.
- [Background] Webb, M. (1999). The Good Death: The New American Search to Reshape the End of Life. New York, Bantam.